CLINICAL TRIAL: NCT05043519
Title: Phase I/II Clinical Trial of NP41 Molecular Targeted Fluorescence Imaging for Cranial Nerve Visualization During Neurosurgery
Brief Title: Phase I/II Clinical Trial of NP41 for Cranial Nerve Fluorescence Imaging
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S2021485
Record Dates: First submitted 2021-09-07; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-08

CONDITIONS: Cranial Nerve Injuries
Keywords: Cranial Nerve; Neurosurgery; Fluorescence Imaging; Molecular Probe; NP41
MeSH Terms: conditions — Cranial Nerve Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FAM-NP41 Fluorescence Imaging (Experimental): The patients will be injected with FAM-NP41 preoperatively, and fluorescence imaging of cranial nerves will be evaluated after the craniotomy.
  Interventions: Drug: FAM-NP41

INTERVENTIONS:
Drug: FAM-NP41 — The patients will be injected with FAM-NP41 in one dose intravenously 2 hours prior to the dural incision.

SUMMARY:
Preclinical evidence has shown that NP41 is a novel nerve-binding peptide with safe pharmacokinetics. Fluorescently labeled NP41 is effective for the intraoperative visualization of cranial nerves during neurosurgery. This Phase I/II clinical trial is aimed to investigate the safety and validity of FAM-NP41 for the fluorescence imaging of cranial nerves. In the Phase I trial, biological safety and adverse events will be evaluated, and pharmacokinetic parameters will be measured. In the Phase II trial, the sensitivity and specificity of FAM-NP41 for the fluorescence imaging of cranial nerves will be investigated, and the signal-to-background ratio will be calculated.

ELIGIBILITY:
Inclusion Criteria:

1. Enhanced brain MRI with or without cranial CT confirms a diagnosis of tumor in the anterior skull base, the middle cranial fossa, or the posterior cranial fossa. Structural images, DTI sequences and 3D-CISS sequences confirm that the tumor is adjacent to the cranial nerve or the cranial nerve will be exposed during the neurological surgery.
2. The body weight is within ±20% of standard body weight [0.7×(height cm-80)]kg;
3. The preoperative laboratory examination parameters of heart, lung, liver, kidney and blood are all in the normal range;
4. Be able to understand the potential risks and benefits of the clinical trial, and sign a written informed consent.

Exclusion Criteria:

1. Preoperative hepatorenal insufficiency: ALT or AST increased ≥ 2 times than the upper limit of normal range; serum creatinine > 2.0 mg/ dL (177 μmol/L) or glomerular filtration rate > 30 ml/min×1.73 m2;
2. Positive reaction in the allergy test, or allergic constitution (such as allergic to two or more foods/drugs, or known to be allergic to protein or to this polypeptide);
3. Preoperative imaging data (enhanced MRI) are incomplete;
4. Serious primary diseases involving important organs;
5. Mentally or physically disabled patients;
6. Alcohol abuse or long-term medication may affect the drug metabolism;
7. According to the judgment of the investigator, the potential intolerance to the drug (such as weak or severe malnutrition);
8. Primary or secondary cranial nerve dysfunction, such as facial paralysis, hearing loss caused by otitis media, etc.
9. Female patients undergoing neurosurgery during pregnancy or lactation.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | 0~24 hours after the drug administration
  Half-life for distribution, half-life for elimination
Hepatorenal functions | 0~72 hours after the drug administration
  ALT, AST, BUN, Cr, GFR
Effectiveness for cranial nerve imaging | Intraoperative period with cranial nerve exposure
  Sensitivity, specificity, signal-to-background ratio

SECONDARY OUTCOMES:
Adverse events | 0~72 hours after the drug administration
  Allergic reaction, changes in vital signs
Functions of cranial nerves | 0~1 week after the drug administration
  Physical examination of cranial nerves

IPD SHARING:
Plan to Share IPD: No